CLINICAL TRIAL: NCT04561310
Title: Comparison of Post Facilitation Stretch and Active Release Technique in Adhesive Capsulitis in Diabetic Patients
Brief Title: Comparison of PFS and ART in Adhesive Capsulitis in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00241 Ummal Baneen
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-09

CONDITIONS: Adhesive Capsulitis
Keywords: Shoulder; Pain; Fibrosis; Disability
MeSH Terms: conditions — Bursitis; Pain; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post facilitation stretch (Experimental): Post facilitation stretch with Maitland mobilization
  Interventions: Other: Post facilitation stretch
- Active release technique (Active Comparator): Active release technique with Maitland mobilization
  Interventions: Other: Active release technique

INTERVENTIONS:
Other: Post facilitation stretch — Post facilitation stretch with maitland mobilization Grade I & II Maitland mobilization of shoulder joint in 1st and 2nd week progressing to Grade III oscillatory mobilization of shoulder joint in 3rd week. It will further progress to Grade IV Maitland oscillatory mobilizations in the 4th or 5th week.
  Treatment will be provided 3 session/week for 6 weeks with 40 minutes/session
  Arms: Post facilitation stretch
Other: Active release technique — Active release technique with maitland mobilization Grade I & II Maitland mobilization of shoulder joint in 1st and 2nd week progressing to Grade III oscillatory mobilization of shoulder joint in 3rd week. It will further progress to Grade IV Maitland oscillatory mobilizations in the 4th or 5th week.
  Treatment will be provided 3 session/week for 6 weeks with 40 minutes/session
  Arms: Active release technique

SUMMARY:
To determine the technique that will have better effects in realigning the muscle kinematics and to normalize the muscle activity along with reducing muscle stiffness with mobilizations techniques

DETAILED DESCRIPTION:
There is a very limited literature available Active release technique (ART) and Post Facilitation Stretch (PFS) in frozen shoulder. Additionally there is a very limited literature on the evaluation of ART in comparison with PFS in adhesive capsulitis of diabetic patient. Disease such as rheumatoid arthritis (RA), osteoarthritis (OA) etc that cause stiffness of the shoulder joint also present with altered muscle activity, that in long run becomes one of the main causes of reduces joint range of motion. With this study, we will be able to determine the technique that will have better effects in realigning the muscle kinematics and to normalize the muscle activity along with reducing muscle stiffness with mobilizations techniques. This study will also fulfill that research gap and will provide clinicians with an alternative approach in treatment of adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Controlled diabetic patients (random 200-250mg/dl /fasting 120-160mg/dl).
* Grade 2 & 3 of adhesive capsulitis,
* Pain (NPRS) ranging between 3-10
* Reduced normal shoulder ROM's i.e

  * Flexion less than 160 degrees.
  * Extension less than 50 degrees.
  * Abduction less than 170 degrees.
  * External rotation less than 80 degrees.
  * Internal rotation less than 70 degrees

Exclusion Criteria:

* Trauma history of shoulder/surgery.
* Frozen shoulder accompanied with neurological involvement.
* People with any injury or disability of elbow or hand

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Shoulder pain and disability Index (SPADI) | 6th week
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.
  Each of the 13 items is to be rated with a number from 0 to 10: For the pain score (first 5 items): 0 means no pain and 10 means worst pain imaginable; For the disability score (last 8 items): 0 means no impairment and 10 means the patient requires help to perform that action
The oxford scale | 6th week
  The Oxford Scale is a 0-5 scale which is then recorded as 0/5 or 2/5, sometimes with a + or - sign to indicate more or less power but not sufficient to reduce or increase the number.
Numeric Pain Rating Scale (NPRS) | 6th week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes.
ROM Shoulder Flexion | 6th week
  Goniometer is used to measure the range of the motion of the shoulder flexion
ROM Shoulder Extension | 6th week
  Goniometer is used to measure the range of the motion of the shoulder extension
ROM Shoulder Abduction | 6th week
  Goniometer is used to measure the range of the motion of the shoulder Abduction
ROM Shoulder External Rotation | 6th week
  Goniometer is used to measure the range of the motion of the shoulder External Rotation
ROM Shoulder Internal Rotation | 6th week
  Goniometer is used to measure the range of the motion of the shoulder Internal Rotation

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Asif Hospital Wah Cantt, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose PG. Effective Reduction of Adhesive Capsulitis Pain with a Suprascapular Nerve Block Given in a Primary Care Clinic. InConference Highlights (p. 30).
- [Background] Ewald A. Adhesive capsulitis: a review. Am Fam Physician. 2011 Feb 15;83(4):417-22. PMID 21322517
- [Background] Tighe CB, Oakley WS Jr. The prevalence of a diabetic condition and adhesive capsulitis of the shoulder. South Med J. 2008 Jun;101(6):591-5. doi: 10.1097/SMJ.0b013e3181705d39. PMID 18475240
- [Background] Garcilazo C, Cavallasca JA, Musuruana JL. Shoulder manifestations of diabetes mellitus. Curr Diabetes Rev. 2010 Sep;6(5):334-40. doi: 10.2174/157339910793360824. PMID 20701586
- [Background] Hsu CL, Sheu WH. Diabetes and shoulder disorders. J Diabetes Investig. 2016 Sep;7(5):649-51. doi: 10.1111/jdi.12491. Epub 2016 Mar 16. No abstract available. PMID 27182002
- [Background] Donatelli R, Ruivo RM, Thurner M, Ibrahim MI. New concepts in restoring shoulder elevation in a stiff and painful shoulder patient. Phys Ther Sport. 2014 Feb;15(1):3-14. doi: 10.1016/j.ptsp.2013.11.001. Epub 2013 Nov 16. PMID 24315683
- [Background] Anton HA. Frozen shoulder. Can Fam Physician. 1993 Aug;39:1773-8. PMID 8374364
- [Background] Gutierrez Espinoza HJ, Pavez F, Guajardo C, Acosta M. Glenohumeral posterior mobilization versus conventional physiotherapy for primary adhesive capsulitis: a randomized clinical trial. Medwave. 2015 Sep 22;15(8):e6267. doi: 10.5867/medwave.2015.08.6267. English, Spanish. PMID 26485477
- [Background] Ravichandran H, Balamurugan J. Effect of proprioceptive neuromuscular facilitation stretch and muscle energy technique in the management of adhesive capsulitis of the shoulder. Saudi Journal of Sports Medicine. 2015 May 1;15(2):170.
- [Background] Vermeulen HM, Rozing PM, Obermann WR, le Cessie S, Vliet Vlieland TP. Comparison of high-grade and low-grade mobilization techniques in the management of adhesive capsulitis of the shoulder: randomized controlled trial. Phys Ther. 2006 Mar;86(3):355-68. PMID 16506872
- [Background] Gupta S, Jaiswal P, Chhabra D. A comparative study between postisometric relaxation and isometric exercises in non-specific neck pain. Journal of exercise science and physiotherapy. 2008;4(2):88.
- [Background] Kim JH, Lee HS, Park SW. Effects of the active release technique on pain and range of motion of patients with chronic neck pain. J Phys Ther Sci. 2015 Aug;27(8):2461-4. doi: 10.1589/jpts.27.2461. Epub 2015 Aug 21. PMID 26357426
- [Background] Shih YF, Liao PW, Lee CS. The immediate effect of muscle release intervention on muscle activity and shoulder kinematics in patients with frozen shoulder: a cross-sectional, exploratory study. BMC Musculoskelet Disord. 2017 Nov 28;18(1):499. doi: 10.1186/s12891-017-1867-8. PMID 29183307
- [Background] Noten S, Meeus M, Stassijns G, Van Glabbeek F, Verborgt O, Struyf F. Efficacy of Different Types of Mobilization Techniques in Patients With Primary Adhesive Capsulitis of the Shoulder: A Systematic Review. Arch Phys Med Rehabil. 2016 May;97(5):815-25. doi: 10.1016/j.apmr.2015.07.025. Epub 2015 Aug 15. PMID 26284892
- [Background] Hung CJ, Hsieh CL, Yang PL, Lin JJ. Relationships between posterior shoulder muscle stiffness and rotation in patients with stiff shoulder. J Rehabil Med. 2010 Mar;42(3):216-20. doi: 10.2340/16501977-0504. PMID 20411215